CLINICAL TRIAL: NCT01205555
Title: Combining Urinary Luteinizing Hormone Testing With Ultrasound Monitoring in Intrauterine Insemination Cycles
Brief Title: Combining LHu With Ultrasound Monitoring in IUI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sufficient participants for analysis
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F-GYN-10-02
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Infertility
Keywords: intra uterine insemination
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound alone group (No Intervention): Patients in the control group will have a standard ultrasound monitoring with HCG administered when the leading follicle reaches 18 mm, and IUI 36 h afterward.
- LH testing combined with ultrasound monitoring (Experimental)
  Interventions: Device: urine LH testing

INTERVENTIONS:
Device: urine LH testing — The study group will start urine LH (LHu) testing according to the mean diameter of the leading follicle on ultrasound as per :
  13mm or less - Repeat ultrasound scan in 1-2 days 14-17mm - start urine LH testing the evening of the day of the scan 18mm or greater - do one LHu test in the afternoon of the day of the scan before HCG administration Once the patient has commenced LHu testing she will perform 2 tests per day. The tests will be performed at 7am and 7pm. LHu testing will continue until the time of HCG administration or positive uLH.If the LHu result is positive either in the morning or afternoon, the insemination will be the next morning without the administration of exogenous HCG.
  If the patient has an inconclusive LHu result, a blood LH test will be taken. If the LH blood test is negative (<8 IU\L) she will continue testing LHu. If the LH blood test is positive (≥ 8 IU\L) the insemination will be the next day.
  Other Names: Conceive Ovulation predictor
  Arms: LH testing combined with ultrasound monitoring

SUMMARY:
Intra-uterine insemination (IUI), generally in combination with ovarian stimulation, is one of the most commonly used treatments for infertility. Accurate timing of insemination, in order to coincide with ovulation, has an important impact on the success rate. Optimal timing of insemination is achieved either by monitoring follicular growth through serial ultrasound measurements followed by the administration of human chorionic gonadotropin (hCG) or by the detection of urinary luteinizing hormone (LH). However in cycles where follicular growth is monitored there is a possibility of premature LH rise before the administration of hCG, which may affect the outcome of the treatment. The goal of the study is to determine if adding the testing of urine LH in conjunction with ultrasound monitoring leads to an increase in pregnancy rates in IUI cycles when compared to ultrasound monitoring alone.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing IUI treatments for:

  * Unexplained infertility (including endometriosis stage 1-2)
  * Mild male factor (>5x106/ml motile sperm as determined by total sperm concentration x % A+B motility in the latest spermogram)
  * Donor insemination
* Natural or stimulated cycles with clomiphene citrate or letrozole
* At least 1 patent tube on hysterosalpingogram, hysterosonogram or laparoscopy within the last two years
* Antral follicular count ≥10 and FSH<10

Exclusion Criteria:

* Polycystic ovarian syndrome or any cause of oligo or anovulation
* Patients taking other infertility medication (metformin, 17B estradiol, progesterone or gonadotropins)
* Presence of an ovarian cyst or a follicle >20 mm on the first ultrasound or any reason for immediate HCG administration
* A previous sperm washing result with less than 5x106/ml motile sperm
* Previous inconclusive uLH test or inability to perform uLH testing

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 367 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 14 days post IUI
  as defined by positive urine pregnancy test

SECONDARY OUTCOMES:
rate of positive LH testing | before hCG administration

CONTACTS AND LOCATIONS:
Overall Officials: Roland Antaki, MD, Principal Investigator — ovo fertilité; Louise Lapensee, MD, Study Director — ovo fertilité; Isaac Jacques Kadoch, MD, Study Director — ovo fertilité; Nicola Dean, PhD, Study Director — ovo fertilité
Locations (1):
- Ovo Fertilité, Montreal, Quebec, Canada